CLINICAL TRIAL: NCT06795659
Title: Combining Esketamine and Prolonged Exposure for PTSD: A Proof-of-Concept Clinical Trial
Brief Title: Combining Esketamine and Prolonged Exposure Treatment for PTSD (Post Traumatic Stress Disorder)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Institute for Integration of Medicine & Science-UT Health San Antonio (Unknown)
Responsible Party: Principal Investigator, Casey Straud, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001076
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: Massed Prolonged Exposure; Esketamine
MeSH Terms: conditions — Combat Disorders | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: Open-label, proof-of-concept, pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Esketamine combined with Prolonged Exposure for PTSD (Experimental): Esketamine (intranasal ketamine) will be administered 6 times over a 2-week period after administering PE sessions
  Interventions: Drug: Esketamine (Intranasal Spray); Behavioral: Massed Prolonged Exposure (PE)

INTERVENTIONS:
Drug: Esketamine (Intranasal Spray) — Esketamine doses will be administered via insufflation with a starting dose of 1 spray of 14 mg per nostril (28 mg/total). Based on tolerability, total dose will be increased to a target dose of 84 mg delivered as three bouts separated by 5 minutes per bout (total dose administered in 15 minutes).
Behavioral: Massed Prolonged Exposure (PE) — Eligible participants will be enrolled to receive 10 sessions of PE delivered in massed (daily) format over 2 weeks (weekdays, not including weekends and holidays)

SUMMARY:
This study is being done to see if Prolonged Exposure (PE), a well-researched, very effective individual (one-to-one) behavioral therapy designed to help people to directly deal with traumatic events they have suffered in the past, can be combined with intranasal esketamine (ketamine) for the treatment of posttraumatic stress disorder (PTSD) to enhance treatment benefits. Ketamine nasal spray is a drug approved by the U.S. Food & Drug Administration (FDA) for treatment resistant depression. Combined with PE, intranasal ketamine may help to augment PE and further reduce participants' PTSD symptoms.

DETAILED DESCRIPTION:
The study is an early phase II, open label, proof of concept, pilot clinical trial to explore the feasibility, acceptability, and effects of esketamine combined with PE in individuals seeking treatment for PTSD. All individuals will complete a phone screen to learn more about the study to discuss broad eligibility criteria. Study candidates will be recruited from provider referrals across the San Antonio community as well as from self-referrals. Interested individuals who appear to meet initial eligibility will be consented and the complete a baseline assessment to determine study eligibility. Eligible participants will be enrolled to receive 10 sessions of PE delivered in massed (daily) format over 2 weeks (weekdays, not including weekends and holidays). Participants will also receive intranasal esketamine six times over a 2-week period (three times a week) approximately 1 hour after PE sessions 1, 3, 5, 6, 8, and 10 over this time period.

ELIGIBILITY:
Inclusion Criteria:

1. Individual between the ages of 18-65 years old (Young adults [18 to 24 years old] must not be taking an antidepressant).
2. PTSD diagnosis as assessed by Clinician-Administered Posttraumatic Stress Scale (CAPS-5)
3. Able to speak and read English (due to standardization of outcome measures)
4. On stable doses of current medications for at least 4 weeks
5. Weigh between 50-100 kg (110-220 pounds).

Exclusion Criteria:

1. Young adults (18-24) currently taking any antidepressant.
2. Lifetime history of psychotic disorder or history of significant psychotic symptoms.
3. Lifetime history of manic episode.
4. Moderate or greater severity for alcohol or substance use disorder (DSM-5) in the previous six months.
5. A history of ketamine or phencyclidine abuse.
6. Evidence of a traumatic brain injury severe enough to interfere with comprehension and responding to the baseline screening questionnaires.
7. Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index-Suicidality Subscale and corroborated by a clinical risk assessment by a credentialed provider)
8. Other psychiatric disorders severe enough to warrant designation as the primary disorder as determined by clinician judgment.
9. Current use (with past 4 weeks) of any prohibited concomitant medications
10. Benzodiazepines, other medications, sedatives, acute alcohol use, or recreational drug use that would put patients at risk in the judgment of clinical providers).
11. Planned use of ketamine (i.e., for pain control) or participation in another trauma-focused psychotherapy during the time of the study.
12. Uncontrolled hypertension or tachycardia
13. A history of sensitivity or adverse reaction to ketamine or its excipients
14. An unstable medical, cardiovascular, pulmonary, or neurological condition that the investigator considers a contraindication to ketamine administration
15. Aneurysmal vascular disease (including thoracic and abdominal aorta, intracranial and peripheral arterial vessels) or arteriovenous malformation.
16. Intracerebral hemorrhage.
17. Pregnancy or breastfeeding; women of childbearing potential unwilling to utilize reliable methods of contraception
18. History of nasal surgery or nasal obstructions experienced as an adult.
19. Inability to arrange for assisted transportation on ketamine treatment days due to recommendation that patient not drive for the remainder of the day following a ketamine treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of Treatment using Esketamine and PE | Study start to closing to enrollment (approximately 12 months)
  Number of eligible referrals
Satisfaction with Therapy and Therapist Scale - Revised (STTS-R) | Day 1 to 1 month
  A12-item self-report measure with strong psychometric properties used to assess the patient's satisfaction with the therapy provided and the therapist. Even number items assess satisfaction with therapy and odd number items assess satisfaction with therapist. Scores can range from 12-60. Higher scores are reflective of greater satisfaction. Items are on a 5-point Likert scale that ranges from 1 = "Strong disagree" to 5 = "Strongly Agree'. Additionally, a 13th item provides an independent assessment of the patient's global improvement. The STTS-R will be administered at the final treatment session and at the 1-month follow-up assessments.
Enrollment proportion | Study start to closed to enrollment (approximately 12 months)
  Proportion of eligible participants
Adherence to treatment | Study start to closed to enrollment (approximately 12 months)
  Number of participants that adhered to and completed treatment
CEQ for Esketamine (Expectancy Score) | Day 1 to 1 month
  The esketamine treatment will be rated as credible with positive expected treatment benefits on the Credibility and Expectancy Questionnaire. Responses to four questions are scored using a 9-point Likert scale (1= not at all, 9= extremely). Responses to two of the questions are scored using an 11-point Likert Scale (0% to 100%). The combined responses are used to generate a score for expectancy.
CEQ for Esketamine (Credibility Score) | Day 1 to 1 month
  The esketamine treatment will be rated as credible with positive expected treatment benefits on the Credibility and Expectancy Questionnaire. Responses to four questions are scored using a 9-point Likert scale (1= not at all, 9= extremely). Responses to two of the questions are scored using an 11-point Likert Scale (0% to 100%). The combined responses are used to generate a score for credibility.
CEQ for PE (Credibility score) | Day 1 to 1 month
  The CEQ for PE is a 6-item measure that was designed to assess treatment expectancy and rationale credibility for use in clinical outcomes studies. Responses to four questions are scored using a 9-point Likert scale (1= not at all, 9= extremely). Responses to two of the questions are scored using an 11-point Likert Scale (0% to 100%). The responses are used to generate a score for credibility.
CEQ for PE (Expectancy score) | Day 1 to 1 month
  The CEQ for PE is a 6-item measure that was designed to assess treatment expectancy and rationale credibility for use in clinical outcomes studies. Responses to four questions are scored using a 9-point Likert scale (1= not at all, 9= extremely). Responses to two of the questions are scored using an 11-point Likert Scale (0% to 100%). The responses are used to generate a score for expectancy.
Post Traumatic Stress Disorder (PTSD) (PCL-5) Checklist-5 Change in Score | Baseline to 1 month
  A 20-item self-report measure designed to assess PSTSD symptoms as defined by the DSM-5 and evaluates how much participants have been bothered by these symptoms in the past week (for all assessments during treatment and one week follow-up) or the past month (all other assessment time points) because of a specific life event. Each item of the PCL-5 is scored on a five-point scale ranging from 0 ("Not at all") to 4 ("Extremely). Scores can range from 0-80. Scores ≥ 33 indicate clinically elevated PTSD symptoms.
The Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (CAPS-5) | Baseline to 1 month
  The CAPS-5 is a structured interview that assesses the DSM-5 criteria for PTSD. Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/Incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Additional items evaluate overall symptom duration, distress, impairment, dissociative symptoms, and global ratings by the interviewer. Subscale scores are calculated by summing severity scores for items in the following PTSD symptom clusters: re-experiencing, avoidance, negative alterations in cognitions and mood, and hyperarousal. Scores ≥ 25 indicate a probable diagnosis of PTSD.

SECONDARY OUTCOMES:
Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Baseline to 1 month
  The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide. Scores on each item range from 0 to 3, with higher scores reflecting greater severity of suicidal ideation. Possible range of scores is from 0-36.
Generalized Anxiety Disorder Screener | Baseline to 1 month
  This is a 7-item measure that asks participants to rate the frequency with which they have been bothered by anxiety symptoms within the past 2 weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Possible scores range from 0-21. Scores on all items are summed to obtain a total severity score. Scores reflect no significant anxiety symptoms (0-4), mild anxiety symptoms (5-9), moderate anxiety symptoms (10-14), and severe anxiety symptoms (>15).
Patient Health Questionnaire-9 | Baseline to 1 month
  It consists of 9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the diagnostic criteria for Major Depressive Disorder. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past 2 weeks (baseline and 1-month follow-up) or 1 week (during treatment and 1-week follow-up) on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores on all items are summed to obtain a total severity score. Scores range from 0-27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (>19).
Posttraumatic Cognitions Inventory (PTCI) | Baseline to 1 month
  The PTCI is a 36-item self-report questionnaire that measures trauma-related thoughts and beliefs. Participants rate their agreement or disagreement with each statement on a 7-point scale, with 1 meaning "totally disagree" and 7 meaning "totally agree". Higher scores indicate a greater endorsement of negative posttraumatic cognitions. Scores range from 36-252.
  The PTCI has three subscales:
  Negative Cognitions of the Self: 21 items (7-63 possible range of score) Negative Cognitions of the World: 7 items (7-49 possible range of score) Self-Blame for the traumatic event: 5 items (7-35 possible range of score)
Brief Inventory of Psychosocial Functioning | Baseline to 1 month
  A 7-item self-report instrument measuring respondents' level of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. Respondents indicate the degree to which they had trouble in the last 30 days in each area on a 7-point scale ranging from 0 ("Not at all") to 6 ("Very much"). Possible scores range from 0-42, with a higher score indicating better psychosocial functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Straud, PsyD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Presentations and publications produced as a result of this work will follow the STRONG STAR Standard Operating Procedure (STRONG STAR-ADM-001-5.0) for Review and Approval of Publications and Presentation and the International Committee of Medical Journal Editors (ICMJE) "Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals" updated January 2024.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion when data are published in a peer review journal.
Access Criteria: At study completion, data will be published in a peer review journal. Any information that is not presented in the publication may be requested through the corresponding author or the STRONG STAR Consortium Repository
URL: https://www.strongstar.org/research/strongstar/strong-star-repository/